CLINICAL TRIAL: NCT00725634
Title: A Phase 1 Study of AV-299 (Formerly SCH 900105) Administered by IV Infusion as Monotherapy in Advanced Solid Tumors, Lymphomas, or Multiple Myeloma or in Combination With Erlotinib in Advanced Solid Tumors
Brief Title: A Phase 1 Dose-Escalation Study in Advanced Solid Tumors, Lymphomas or Multiple Myeloma
Acronym: P05538
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05538
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Malignant Solid Tumor; Lymphomas; Multiple Myeloma
Keywords: Neoplasms,; Lymphoma,; Multiple Myeloma,; Neoplasms, Plasma Cell,; Neoplasms by Histologic Type,; Lymphoproliferative Disorders,; Lymphatic Diseases, Immunoproliferative Disorders; Immune System Diseases Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Erlotinib; Protein Kinase Inhibitors; Enzyme Inhibitors,; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders | interventions — ficlatuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AV-299 Dose Escalation Arm (Experimental): AV-299 Administered by IV Infusion as Monotherapy in Advanced Solid Tumors, Lymphomas, or Multiple Myeloma
  Interventions: Biological: AV-299
- AV-299 in combination with erlotinib (Experimental): AV-299 Administered by IV Infusion in Combination with Erlotinib (150 mg daily) in Advanced Solid Tumors
  Interventions: Biological: AV-299 + erlotinib

INTERVENTIONS:
Biological: AV-299 — AV-299 monotherapy will be given as intravenous infusion in dose-escalation cohorts at 2, 5, 10, and 20 mg/kg. Once the RP2D has been determined the cohort may be expanded to include up to 12 patients for safety assessment and enriched with up to 12 additional Multiple Myeloma patients.
  Other Names: Formerly SCH 900105
  Arms: AV-299 Dose Escalation Arm
Biological: AV-299 + erlotinib — AV-299 will be given as intravenous infusion at RP2D in combination with erlotinib (150 mg daily). Once the combination-RP2D has been determined the cohort may be expanded to include up to 12 additional patients.
  Other Names: Formerly SCH 900105
  Arms: AV-299 in combination with erlotinib

SUMMARY:
Phase 1 study to determine safety, tolerability, dose-limiting toxicities (DLTs), and recommended Phase 2 dose of AV-299 administered IV as monotherapy to patients with relapsed or refractory solid tumors, lymphoma, or multiple myeloma. The study will also determine the safety, tolerability and DLTs of AV-299 in combination with erlotinib in patients with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an advanced solid tumor malignancy or lymphoma (non-Hodgkin's or Hodgkin's lymphoma).
* Histological or cytological evidence of malignancy.
* Advanced malignancy, metastatic or unresectable, that has recurred or progressed following standard therapy or failed standard therapy; or for which no standard therapy currently exists, or for which subject is not a candidate for, or is unwilling to undergo, standard therapy.
* Disease that is currently not amenable to curative surgical intervention.
* ECOG performance status of 0-1. Subjects with performance status of 2 will be considered only after discussion between the investigator and medical monitor.
* 18 years or older, of either sex, and of any race.
* Subject (and/or parent/guardian for subject who otherwise is unable to provide independent consent, if acceptable to and approved by the site and/or site's IRB) must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Female subjects of childbearing potential must have negative pregnancy test within 5 days prior to first dose of study drug.
* Female subjects of childbearing potential and male subjects whose sexual partners are of childbearing potential must agree to abstain from sexual intercourse or to use an effective method of contraception during the study and for 60 days after the last dose of AV-299 (formerly SCH 900105). Examples of effective methods of contraception include, but are not limited to, oral contraceptives or double barrier methods such as condom plus spermicide or condom plus diaphragm.
* Adequate hematologic function as evidenced by Hg ≥ 9g/dL, WBC ≥ 3000 per mm3, ANC ≥ 1500 per mm3 and platelet count ≥ 100,000 per mm3.
* Adequate hepatic function as evidenced by a serum bilirubin level ≤1.5 × ULN (except with known Gilbert's Syndrome) and
* For subjects in the dose-escalation cohorts and the Phase 1b evaluation of AV-299 (formerly SCH 900105) in combination with erlotinib:

  -- Serum AST/ALT levels ≤3 × ULN for the reference laboratory
* For subjects in the RP2D safety expansion cohort:

  * Without known hepatic metastasis serum AST/ALT levels ≤3 × ULN for the reference laboratory
  * With known hepatic metastasis serum AST/ALT levels ≤5 × ULN.
  * Adequate renal function as evidenced by a serum creatinine level ≤ 1.5 × ULN or a calculated creatinine clearance > 60 mL/min.
  * Adequate coagulation function as evidenced by PTT ≤ 1.5 × ULN and INR ≤ 1.5 × ULN
  * Recovery from the effects of any prior surgery, radiotherapy, or systemic antineoplastic therapy.
  * Subjects with abnormal liver function tests (LFTs) who have not been screened for Hepatitis B or C within the past 6 months prior to study enrollment, will need to be screened for Hepatitis B and C and can only be enrolled if the screening is negative.

Diagnosis and Main Criteria for Inclusion for the Multiple Myeloma Exploratory Cohort Subjects to be Included

* Diagnosis of symptomatic relapsed or refractory multiple myeloma. Note: For relapsed disease, subject must have PD after having achieved at least stable disease for ≥ 1 cycle of treatment to ≥ 1 prior regimen. For refractory disease, subject must have documented evidence of PD during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry.
* Measurable disease assessed by one of the following:

  * Serum monoclonal protein ≥ 1.0 g/dL by protein electrophoresis;
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis;
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio; or,
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease). Note: All above evaluations, for which there are measurable results at screening, will be repeated as indicated in the visit schedule and the schedule of assessments, with the exception of bone marrow plasmacytosis. Bone marrow plasmacytosis will be repeated for disease/response assessment according to the visit schedule and the schedule of assessments if it is the only measurable result at screening. If both serum and urine M-proteins are present, both must be followed in order to evaluate response.
* At least 2 prior therapies
* ECOG performance status of 0, 1, or 2.
* 18 years or older, of either sex, and of any race.
* Subject (and/or parent/guardian for subject who otherwise is unable to provide independent consent, if acceptable to and approved by the site and/or site's IRB) must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Female subjects of childbearing potential must have negative pregnancy test within 5 days prior to first dose of study drug.
* Female subjects of childbearing potential and male subjects whose sexual partners are of childbearing potential must agree to abstain from sexual intercourse or to use an effective method of contraception during the study and for 60 days after the last dose of AV-299 (formerly SCH 900105). Examples of effective methods of contraception include, but are not limited to, oral contraceptives or double barrier methods such as condom plus spermicide or condom plus diaphragm.
* Adequate hematologic function as evidenced by Hg ≥ 9g/dL, ANC ≥ 1000 per mm3, and platelet count ≥ 50,000 per mm3. Screening platelet count should be independent of platelet transfusions for ≥ 2 weeks.
* Adequate hepatic function as evidenced by a serum bilirubin level ≤ 1.5 × ULN (except with known Gilbert's Syndrome) and serum AST and ALT levels ≤ 3 × ULN.
* Adequate renal function as evidenced by a serum creatinine level ≤ 3.0 mg/dL.
* Adequate coagulation function as evidenced by PTT ≤ 1.5 × ULN and INR ≤ 1.5 × ULN.
* All previous cancer chemotherapy, including radiation, hormonal therapy, and surgery, must have been discontinued ≥ 2 weeks prior to first dose of study drug.
* Subjects with abnormal liver function tests (LFTs) who have not been screened for Hepatitis B or C within the past 6 months prior to study enrollment, will need to be screened for Hepatitis B and C and can only be enrolled if the screening is negative.
* Subject willing to provide blood and if feasible, bone marrow samples for research purposes.

Exclusion Criteria:

* Women who are breast-feeding, pregnant, or intend to become pregnant.
* Subjects with primary CNS malignancy or symptomatic CNS metastases, with the exception that subjects with glioblastoma multiforme may be enrolled in the RP2D Safety Expansion Cohort and in the Phase 1b evaluation of AV-299 (formerly SCH 900105) in combination with erlotinib. Subjects with treated brain metastases that have remained stable for at least 3 months without steroids are allowed. Subjects with signs or symptoms or history of brain metastasis must have a CT or MRI scan of the brain within 1 month prior to the first dose of study drug. Subjects with spinal cord or nerve root compression who have completed treatment at least 4 weeks prior to the first dose of study drug and are stable without steroid treatment for at least 1 week prior to the first dose of study drug are allowed. Subjects with leptomeningeal metastases are not allowed.
* Hematologic malignancies other than lymphoma
* Any of the following within 6 months prior to administration of study drug:

Myocardial infarction (MI), severe /unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or seizure disorder.

* Serious and/or symptomatic active infection within 14 days prior to first dose of study drug. Subjects who have asymptomatic or mild infection and taking a short course of antibiotics (ie, UTI, bronchitis) may be allowed after discussion with the medical monitor.
* Baseline QTc interval as follows per Bazett's formula: Females > 470 msec; Males > 450 msec.
* Persistent, unresolved CTCAE v3.0 Grade 2 or higher drug-related toxicity (except alopecia, erectile dysfunction, hot flashes, and decreased libido) associated with previous treatment.
* Inadequate recovery from any prior surgical procedure or major surgical procedure performed within 4 weeks prior to administration of first dose or major surgery within 3 weeks prior to first dose of study drug.
* Any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* Known Human Immunodeficiency Virus (HIV) infection or a known HIV-related malignancy.
* Known active hepatitis B or C.
* Known hypersensitivity to any of the components of AV-299 (formerly SCH 900105).
* Radiotherapy within 3 weeks prior to first study drug administration.
* Inability to comply with the protocol requirements or participation in any other clinical study.
* Any medications listed in the table on "Prohibited Medications".
* Active alcohol abuse.
* Stem cell/bone marrow transplant within 6 months of first dose of study drug.

Additional Exclusion Criteria for Subjects Enrolled in the Phase 1b Evaluation of AV-299 (formerly SCH 900105) in Combination with Erlotinib:

* Inability to take oral medications
* Grade 2 or higher diarrhea at baseline, or inflammatory bowel disease
* Any gastrointestinal disorder that may interfere with the absorption of oral medications
* Acute onset of new or progressive pulmonary symptoms, such as dyspnea, cough or fever within 4 weeks prior to first study treatment, or diagnosis of interstitial lung disease (ILD)

Exclusion for the Multiple Myeloma Exploratory Cohort

* Women who are breast-feeding, pregnant, or intend to become pregnant.
* Active malignancy of any kind requiring or likely to require treatment within the next 12 months, with the exception of basal cell skin cancer, in situ cervical cancer, in situ breast cancer and asymptomatic prostate cancer.
* Any of the following prior to first dose of study drug: POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), plasma cell leukemia, Waldenstrom's macroglobulinemia.
* Any of the following within 6 months prior to administration of study drug:

Myocardial infarction (MI), severe /unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or seizure disorder.

* Serious and/or symptomatic active infection within 14 days prior to first dose of study drug. Subjects who have asymptomatic or mild infection and taking a short course of antibiotics (ie, UTI, bronchitis) may be allowed after discussion with the medical monitor.
* Baseline QTc interval as follows per Bazett's formula: Females > 470 msec; Males > 450 msec.
* Persistent, unresolved CTCAE v3.0 Grade 2 or higher drug-related toxicity (except alopecia, erectile dysfunction, hot flashes, and decreased libido) associated with previous treatment.
* Inadequate recovery from any prior surgical procedure or major surgical procedure performed within 4 weeks prior to administration of first dose or major surgery within 3 weeks prior to first dose of study drug.
* Any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* Known Human Immunodeficiency Virus (HIV) infection or a known HIV-related malignancy.
* Known active hepatitis B or C.
* Known hypersensitivity to any of the components of AV-299 (formerly SCH 900105).
* Radiotherapy within 3 weeks prior to first study drug administration, except when used as palliative treatment for pain control.
* Inability to comply with the protocol requirements or participation in any other clinical study.
* Any medications listed in the table on "Prohibited Medications".
* Active alcohol abuse.
* Maintenance steroid therapies of > 20 mg/day prednisone, > 4 mg/day dexamethasone, > 80 mg/day hydrocortisone, or equivalent.

NOTE: Maintenance steroid therapies of ≤ 20 mg/day prednisone, ≤ 4 mg/day dexamethasone, ≤ 80 mg/day hydrocortisone, or equivalent are allowed provided that the subject is on a stable dose for at least 2 weeks prior to first dose of study drug or the dose has not been adjusted upwards in the 2 weeks prior to first dose of study drug.

* Prior therapy involving anti-HGF antibody or c-Met small molecule inhibitor.
* Allogeneic stem cell/bone marrow transplant within 12 months of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity and Recommended Phase 2 dose | Following 4 weeks of treatment
  Assessment of any dose-limiting toxicity

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of AV-299, and erlotinib (for subjects enrolled in the Phase 1b only). | Cycle 1: Day 1-4, Day 8 Cycle 2: Day 1, Day 8 Cycle 3: Day 1 Cycle 4: Day 8-14 Subsequent Cycles to Cycle 52: Day 1 End of Treatment Visit 1-Month and 2-Month Follow-Up Visits
Evaluate the effects of AV-299 and combination of AV-299 and erlotinib on exploratory biomarkers in blood, body fluid, tumor tissue, and/or bone marrow. | Screening Cycle 1: Day 1-4, Day 8 Cycle 2: Day 1, Day 8-14 Cycle 4: Day 8-14
Study the preliminary antineoplastic activity of AV-299 in subjects with advanced solid tumors, lymphoma, or multiple myeloma, and the preliminary antineoplastic activity of AV 299 in combination with erlotinib in subjects with advanced solid tumor. | Advanced solid tumors and lymphoma, every 8 weeks through Cycle 29, and approximately every 12 weeks thereafter. Subjects with multiple myeloma will undergo disease assessment at screening and approximately every 4 weeks after Day 1.
Investigate the effect of AV-299 and of the combination of AV-299 and erlotinib on gene expression patterns in peripheral blood mononuclear cells and/or bone marrow. | Cycle 1: Day 1-4 Cycle 4: Day 8-14
Assess dosing schedules of AV-299 (e.g. every 2-week and every 3-week schedules). | Throughout the study
Assess safety and tolerability of the RP2D of AV-299 in expansion cohort(s). | Throughout the expansion cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Philip Komarnitsky, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Investigational Site 2, Scottsdale, Arizona
  - Investigational Site 3, Columbus, Ohio
  - Investigational Site 1, San Antonio, Texas